CLINICAL TRIAL: NCT07101536
Title: The Application of mRNA Immunotherapy Technology in Refractory Malignancies Associated With Epstein-Barr Virus (EBV)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBV-mRNA-2025
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: EBV-associated Tumors
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EBV mRNA vaccine, Dose 1 (Experimental)
  Interventions: Biological: EBV mRNA vaccine
- EBV mRNA vaccine, Dose 2 (Experimental)
  Interventions: Biological: EBV mRNA vaccine
- EBV mRNA vaccine, Dose 3 (Experimental)
  Interventions: Biological: EBV mRNA vaccine
- EBV mRNA vaccine, Expanded dose (Experimental)
  Interventions: Biological: EBV mRNA vaccine
- EBV mRNA vaccine, Combination therapy (Experimental)
  Interventions: Biological: EBV mRNA vaccine; Biological: Immune Checkpoint Inhibitors, ICIs

INTERVENTIONS:
Biological: EBV mRNA vaccine — EBV mRNA vaccine
Biological: Immune Checkpoint Inhibitors, ICIs — Immune Checkpoint Inhibitors, ICIs
  Arms: EBV mRNA vaccine, Combination therapy

SUMMARY:
Epstein-Barr virus (EBV) is an important tumor-associated virus. In 1997, the World Health Organization (WHO) officially classified EBV as a Group 1 carcinogen, as it is implicated in the pathogenesis of various epithelial malignancies and multiple types of lymphomas. Epithelial malignancies associated with EBV infection include nasopharyngeal carcinoma (NPC), gastric cancer, colorectal cancer, breast cancer, cervical cancer, prostate cancer, and oral cancer, among others. Currently, optimal therapeutic strategies for EBV-associated tumors remain lacking, particularly in patients with recurrent, metastatic, or refractory disease. Furthermore, although EBV infection plays a significant role in the development and progression of EBV-positive tumors and may influence patient prognosis, there are currently no precision therapeutic approaches specifically targeting EBV-positive lymphomas. Thus, treatment options for this patient population warrant further attention.

EBV mRNA vaccine is a therapeutic vaccine based on messenger RNA (mRNA) targeting antigens related to EBV. This clinical trial aims to evaluate the safety, tolerability, immunogenicity, and preliminary antitumor activity of EBV mRNA vaccine in patients with advanced EBV-positive malignant tumors, thereby providing a scientific basis for subsequent clinical development.

ELIGIBILITY:
Inclusion Criteria:

Phase 1: Monotherapy Study of mRNA Vaccine

* Male or female patients aged ≥18 years;
* Patients with advanced Epstein-Barr virus (EBV)-positive tumors (e.g., nasopharyngeal carcinoma, NK/T-cell lymphoma, or gastric cancer) who have failed at least two lines of standard therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-2;
* Estimated survival ≥3 months;
* Adequate major organ function;
* Additional inclusion criteria may be supplemented.

Phase 2: Combination Therapy Study of mRNA Vaccine

* Male or female patients aged ≥18 years at screening;
* Histopathologically confirmed recurrent or metastatic nasopharyngeal carcinoma (NPC) not amenable to local therapy, with documented failure of at least one prior platinum-containing chemotherapy regimen and PD-1/L1 immunotherapy;
* Positive for Epstein-Barr virus-encoded RNA (EBER) in tumor tissue;
* At least one measurable lesion per RECIST v1.1 criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-2;
* Additional inclusion criteria may be supplemented.

Exclusion Criteria:

Phase 1: Monotherapy Study of mRNA Vaccine

* Participation in another clinical drug trial within the past 4 weeks;
* History of other malignancies, unless it is cervical carcinoma in situ, treated cutaneous squamous cell carcinoma or urothelial tumors, or other malignancies that have undergone curative treatment (at least 5 years prior to enrollment);
* Uncontrolled cardiac symptoms or diseases;
* Female subjects who are pregnant or breastfeeding;
* Active tuberculosis, bacterial or fungal infections; active HIV infection, active HBV infection, or HCV infection;
* Additional exclusion criteria may be supplemented.

Phase 2: Combination Therapy Study of mRNA Vaccine

* History of other primary malignancies within 3 years prior to the first dose, excluding adequately treated tumors with no evidence of recurrence for at least 2 years;
* Known clinically significant uncontrolled cardiac symptoms or diseases;
* Presence of central nervous system disorders (e.g., epilepsy, severe cerebrovascular stenosis), or history of cerebrovascular accident (e.g., stroke) or other cerebrovascular events within 6 months prior to screening, or other conditions (including psychiatric disorders) with overt neurological symptoms;
* Known history of interstitial pneumonia or high suspicion of interstitial pneumonia; or presence of pulmonary abnormalities that may interfere with the detection or management of suspected drug-related pulmonary toxicity during the trial;
* Any active autoimmune disease or history of autoimmune diseases;
* Additional exclusion criteria may be supplemented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During one year after initial treatment
Safety: Type, frequency, and severity of treatment-related adverse events | During one year after initial treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | During one year after initial treatment
Disease control rate (DCR) | During one year after initial treatment
Progression-free survival (PFS) | During one year after initial treatment
Survival rate (1-year, 2-year) | During one and two years after initial treatment

IPD SHARING:
Plan to Share IPD: Undecided